CLINICAL TRIAL: NCT00591344
Title: The Effect of Exercise on Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Daniel Corcos, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NS028127 (NIH); 5R01NS028127-16 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive resistance training (Active Comparator): Subjects will perform between 60 and 90 minutes of progressive resistance training two times a week for two years at a local gym. These sessions will be supervised by a personal trainer two times a week for the first six months of training and then once a week for the remaining 18 months of training.
  Interventions: Behavioral: Progressive resistance training
- Modified Fitness Counts (Active Comparator): Subjects will perform between 60 and 90 minutes of modified Fitness Counts two times a week for two years at a local gym. These sessions will be supervised by a personal trainer two times a week for the first six months of training and then once a week for the remaining 18 months of training.
  Interventions: Behavioral: Modified Fitness Counts

INTERVENTIONS:
Behavioral: Progressive resistance training — Exercise twice a week for 2 years doing either progressive resistance training. The The PRE program consisted of 11 strengthening exercises: chest press, latissimus pull downs, reverse flys, double leg press, hip extension, shoulder press, biceps curl, rotary calf (ankle plantar flexion), triceps extension, seated quadriceps extension and back extension.
  Arms: Progressive resistance training
Behavioral: Modified Fitness Counts — The modified Fitness Counts program was taken from Chapters 2 and 3 of the Parkinson's disease: Fitness Counts booklet and focused on non-progressive stretching, strengthening and balance exercises.
  Arms: Modified Fitness Counts

SUMMARY:
The goal of this trial is to compare the effect of two different exercise programs on neuro-physiological, motor, functional, and quality-of-life issues in individuals with Parkinson's disease to determine which program is most beneficial.

DETAILED DESCRIPTION:
Parkinson's disease (PD) negatively affects the quality of life for a million individuals in the United States. While medication and surgery are the most effective treatments for PD, physicians and people with PD often delay using these treatments because of their considerable adverse side effects. Until a cure for PD is discovered, there is a compelling need to develop interventions that provide relief of symptoms without causing negative side effects.

Recent research suggests that exercise may provide symptom relief in some characteristics of PD. While various exercise interventions appear to effectively improve motor, functional, and quality-of-life issues, the research is mixed regarding the nature, extent and duration of these improvements. Understanding how multiple characteristics of PD change and whether they can be modified by different exercise programs is essential to determining if an exercise program is clinically effective for PD.

This study is designed to compare the initial (six months), and then long-term (2 years) effect that 2 different exercise programs (progressive resistance program or flexibility program) have on neuro-physiological, motor, functional, and quality-of-life issues in individuals with Parkinson's disease. The goal is to determine which program is most beneficial. Results from this study will be used to determine which exercise program produces the most beneficial effects on neuro-physiological, motor, functional and quality-of-life measures.

NOTE: Recruitment for Parkinson's disease participants is now closed.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of PD
* Up to the age of 67
* on at least 1 DA drug, may be on several PD medications
* able to walk for six minutes (may take rest breaks)
* able to come off their PD medication for testing (12 hour overnight withdrawal of antiparkinsonian medications)
* able to stay on stable PD medications for at least 6 months
* live within a 30 mile radius of Chicago
* Hoehn and Yahr Score: II - III while in the "Off" PD medication state

Exclusion Criteria:

* history of any other neurological disorder as determined by medical history and neurological exam
* history of a known injury, disease, or other disorder that might interfere with motor function in the proposed experiments
* a score less than 23 on the Mini-Mental State Examination
* currently involved in an active, ongoing formal exercise program deep brain stimulation surgery
* known cardiac problem or significant hypertension
* depression that may interfere with regular exercise
* hallucinations or being treated for hallucinations

Ages: 50 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-10; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Corcos, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Physical Therapy Department at the University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] David FJ, Robichaud JA, Leurgans SE, Poon C, Kohrt WM, Goldman JG, Comella CL, Vaillancourt DE, Corcos DM. Exercise improves cognition in Parkinson's disease: The PRET-PD randomized, clinical trial. Mov Disord. 2015 Oct;30(12):1657-63. doi: 10.1002/mds.26291. Epub 2015 Jul 6. PMID 26148003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Parkinson's disease, confirmed by a Movement Disorders specialist, were self-referred or recruited from Rush University Medical Center (RUMC) between 9/2007 and 7/2011 for PD subjects. Patients were evaluated at the University of Illinois at Chicago (UIC).
Pre-assignment Details: Patients were 50 to 67 years; on stable PD meds; and can walk for 6 minutes. Patients were ineligible if they had a neurological history other than PD; significant arthritis; failed the Physical Activity Readiness Questionnaire; had cognitive impairment (indicated by Mini-Mental State Examination score); actively exercising; or had surgery for PD.
Groups:
- 1 Progressive Resistance Training: Subjects performed between 60 and 90 minutes of progressive resistance training two times a week for two years at a local gym. These sessions were supervised by a personal trainer two times a week for the first six months of training and then once a week for the remaining 18 months of training.
  Exercises included progressive resistance training. Participants exercised twice a week for 2 years doing progressive resistance training.
- 2 Modified Fitness Counts: Subjects performed between 60 and 90 minutes of flexibility training two times a week for two years at a local gym. These sessions were supervised by a personal trainer two times a week for the first six months of training and then once a week for the remaining 18 months of training.
  Exercise inlcuded flexibility training. Participants exercised twice a week for 2 years doing flexibility training.
Period: Overall Study
Arm/Group | 1 Progressive Resistance Training | 2 Modified Fitness Counts
Started | 25 (25 randomized, 1 withdrew before the 6 month test and was replaced; 24 completed the 6 month test) | 26 (26 randomized, 2 withdrew before the 6 month test and were replaced, 24 completed 6 month test)
Completed the 6 Month Test | 24 (Number of subjects who completed the 6 month test) | 24 (Number of subjects who completed the 6 month test)
Completed | 20 (Number of subjects who completed the final 24 month test) | 18 (Number of subjects who completed the final 24 month test)
Not Completed | 5 | 8
Not completed — Transportation issues | 1 | 0
Not completed — Moved out of state | 1 | 0
Not completed — Medical complications | 1 | 3
Not completed — Underwent DBS | 2 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not want to come off medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 1 Progressive Resistance Training: 25 PD Subjects performed between 60 and 90 minutes of progressive resistance training two times a week for two years at a local gym. These sessions were supervised by a personal trainer two times a week for the first six months of training and then once a week for the remaining 18 months of training.
  Exercises included progressive resistance training. Participants exercised twice a week for 2 years doing progressive resistance training.
- 2 Flexibility Training: 25 PD subjects performed between 60 and 90 minutes of flexibility training two times a week for two years at a local gym. These sessions were supervised by a personal trainer two times a week for the first six months of training and then once a week for the remaining 18 months of training.
  Exercise inlcuded flexibility training. Participants exercised twice a week for 2 years doing flexibility training.
- Total: Total of all reporting groups
Arm/Group | 1 Progressive Resistance Training | 2 Flexibility Training | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (5.6) | 59.0 (4.6) | 58.8 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Off Medication UPDRS Part III, Motor Subscale Score
Description: UPDRS part III, is an observer rated clinical measure of motor signs of PD. It is used as a measure of severity of motor signs. We measured this at baseline, 6 , 18 and 24 months. This is a ordinal scale of 0-4 which has 27 items which measures slowness of movement (Bradykinesia), Tremor, Rigidity (muscle stiffness) and postural instabilty. The total value for UPDRS part III scale which ranges from 0 to 108, with a larger number indicating a higher level of impairment.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Modified Fitness Counts: Baseline Assessment- off medication UPDRS part III, motor subscale score
- Progressive Resistance Exercise: Baseline Assessment - off medication UPDRS part III, motor subscale score
Arm/Group | Modified Fitness Counts | Progressive Resistance Exercise
Number analyzed (Participants) | 24 | 24
units on a scale
  baseline | 34.7 (11.5) | 34.5 (11.9)
  6 month | 29.3 (12.2) | 28.0 (10.9)
  12 month | 32.8 (12.4) | 28.4 (10.8)
  18 month | 32.8 (12.3) | 28.6 (9.4)
  24 month | 34.0 (12.6) | 25.8 (10.6)

2. Secondary Outcome: On Medication UPDRS-III
Description: UPDRS part III, is an observer rated clinical measure of motor signs of PD. It is used as a measure of severity of motor signs. We measured this at baseline, 6 , 18 and 24 months. This is a ordinal scale of 0-4 which has 27 items which measures slowness of movement (Bradykinesia), Tremor, Rigidity (muscle stiffness) and postural instabilty. The total value for the UPDRS part III scale which ranges from 0 to 108, with a larger number indicating a higher level of impairment.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Modified Fitness Counts: Baseline Assessment- on medication UPDRS part III, motor subscale score
- Progressive Resistance Exercise: Baseline Assessment - on medication UPDRS part III, motor subscale score
Arm/Group | Modified Fitness Counts | Progressive Resistance Exercise
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 20.9 (8.0) | 21.6 (10.1)
  6 month | 17.7 (8.6) | 19.1 (9.0)
  12 month | 19.1 (8.4) | 19.4 (8.5)
  18 month | 18.1 (9.7) | 18.4 (6.5)
  24 month | 19.3 (9.7) | 17.9 (8.7)

3. Secondary Outcome: L-dopa equivalent-mg/Day
Description: This was the equivalent amount of dopamine (mg/day) each subject was prescribed based upon all of their PD medications.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Measure: Mean (Standard Deviation); unit: mg/day
Groups:
- Modified Fitness Counts; Progressive Resistance Exercise: Baseline Assessment- L-dopa equilivent-mg/day
Arm/Group | Modified Fitness Counts | Progressive Resistance Exercise
Number analyzed (Participants) | 24 | 24
mg/day
  Baseline | 704.5 (405.3) | 597.8 (355.2)
  6 month | 741.2 (443.5) | 619.0 (370.6)
  12 month | 772.2 (472.7) | 638.1 (352.2)
  18 month | 907.9 (546.9) | 691.4 (384.5)
  24 month | 934.1 (557.2) | 753.6 (369.4)

4. Secondary Outcome: Elbow Flexion Strength
Description: This is the MVC for elbow flexion
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

5. Secondary Outcome: Ankle Plantar Flexion Strength
Description: This is a measure of the MVC for ankle plantar flexion strength
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

6. Secondary Outcome: Elbow Extension Strength
Description: This is a measure of the MVC for elbow extension
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

7. Secondary Outcome: Ankle Dorsiflexion Strength
Description: This is a measure of the MVC for ankle dorsiflexion
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

8. Secondary Outcome: Percentage of Agonist EMG Signal Contained in the 0-5, 5-15, 15-30, and 35-50 Hz Frequency Bins During Isometric Contractions
Description: This is a measure of the percentage of the EMG signal that is contained in different frequency bins during a MVC (elbow flexion/extension; ankle DF/PF), a 50% of MVC elbow fleixon contraction, and a 5 NM elbow flexion contraction.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

9. Secondary Outcome: The Integral of the First Agonist Burst
Description: The Integral of the first agonist EMG signal from onset of the agonist EMG signal until peak velocity
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

10. Secondary Outcome: Magnitude of the First 30 ms of the Agonist Burst
Description: The integral of the first 30 msec of the agonist EMG.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

11. Secondary Outcome: Magnitude of the Antagonist Burst
Description: the area under the rectified antagonist signal form agonist EMG onset until the end of movement. This reflects the amount of antagonist activation during movement.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

12. Secondary Outcome: Magnitude of the Agonist Burst
Description: Magnitude of the agonist burst reflects the amount of agonist activation during movement.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

13. Secondary Outcome: Duration of First Agonist Burst
Description: Time in (ms) for the duration of the first agonist burst during a 72 degree elbow flexion movement and also the percentage of agonist EMG bursts until peak velocity
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

14. Secondary Outcome: Number of Agonist Bursts
Description: This is the number of agonist bursts prior to peak velocity.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

15. Secondary Outcome: Co-contraction During Limb Acceleration
Description: the amount of agonist and antagonist activity present during limb acceleration.
Time Frame: Obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

16. Secondary Outcome: Qant
Description: The integral of the antagonist EMG signal from the onset of the agonist EMG to the end of the movement
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

17. Secondary Outcome: Time to Peak Velocity
Description: Time of the onset of the movement to peak velocity.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

18. Secondary Outcome: Peak Movement Velocity
Description: This is how fast an individual can perform a 72 degree elbow flexion movement
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

19. Secondary Outcome: Relaxation Time
Description: Time for a subject to passively relax their muscle after performing and isometric contraction to 50% of their MVC
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

20. Secondary Outcome: Rise Time
Description: This is the time is takes for an individual to go for rest to a 50% of a MVC contraction as fast as possible.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

21. Secondary Outcome: Spatiotemporal Gait Analysis
Description: Spatiotemporal gait analysis using a pressure sensitive walk way allow for measurement of gait velocity, step length, single and double limb support time, cadence, ect.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

22. Secondary Outcome: Distance Walked in 6 Minutes
Description: This is how far an individual can walk in 6 minutes
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

23. Secondary Outcome: Modified Physical Performance Test
Description: This is an overall measure of physical fuction
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

24. Secondary Outcome: Time on the Timed up and go Test
Description: This is the time it takes an individual to get up from a chair, walk 3 meters, turn around and walk back.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

25. Secondary Outcome: Berg Balance Scale Score
Description: This is a overall measure of balance
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

26. Secondary Outcome: Functional Reach
Description: The distance one can reach forward without taking a step.
Time Frame: Obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

27. Secondary Outcome: Cognitive Function - Stroop Test
Description: This is a test of cognitive function. This test requires individuals to first say as many colors as they can under three different test conditions.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

28. Secondary Outcome: Cognitive Function - Brief Test of Attention
Description: This is a cognitive test of an individuals ability to remember number. It is a test of working memory.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

29. Secondary Outcome: Cognitive Function - Digit Span Forward/Backward
Description: This tests a persons ability to remember that were read to them both forward and then backwards.
Time Frame: obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

30. Secondary Outcome: Parkinson 's Disease Quality of Life
Description: PDQ-39 is a composite measure of quality of life in individuals with Parkinson's Disease.
Time Frame: Obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

31. Secondary Outcome: Epworth Sleepiness Scale
Description: The Epworth Sleepiness Scale is used to determine the level of daytime sleepiness.
Time Frame: Obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

32. Secondary Outcome: Beck's Depression Inventory
Description: This is a self-report rating inventory that measures characteristic attitudes and symptoms of depression.
Time Frame: Obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

33. Secondary Outcome: 50 ft Walk Time
Description: Time it takes to walk 50 feet
Time Frame: Obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

34. Secondary Outcome: 50 Foot Walk Speed
Description: The speed that aerson walks over 50 feet
Time Frame: Obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

35. Secondary Outcome: 5 Time Sit to Stand
Description: The time it takes to stand up and sit down five times
Time Frame: Obtained during initial evaluation & then every 6 six months to end of 2-yr training period
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: SAE's and AE's were collected for 2 years for each study participant.
Arm/Group | 1 Progressive Resistance Training | 2 Modified Fitness Counts
Serious Adverse Events (participants affected / at risk) | 8/25 | 6/26
Other Adverse Events (participants affected / at risk) | 0/25 | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Progressive Resistance Training (N=25) | 2 Modified Fitness Counts (N=26)
Passed away (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Passed away after getting hit by a car
DBS surgery (Nervous system disorders) | 2 (2) | 2 (2)
ALS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Developed ALS during the study
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Hospitalization for bowel obstruction
Elbow pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Occurred after fall at home and required medical intervention
Back surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Back surgery for stenosis
Bilateral hip replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
unilateral knee replacement (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) — Pt had both knees replaced during separate surgeries
Knee surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Knee surgery to remove old debris
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Long term hospitalization after fall at home
Foot surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Progressive Resistance Training (N=25) | 2 Modified Fitness Counts (N=26)
Wrist pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Wrist pain while during MVC during testing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No